CLINICAL TRIAL: NCT06969469
Title: To Evaluate the Influence of (LUA Probiotics) on Uric Acid
Status: Completed | Type: Observational
Sponsor: Grape King Bio Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Grape King Bio Ltd
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hyperuricemia (uric acid level 7.5 mg/dL or above): Patients with hyperuricemia (uric acid level 7.5 mg/dL or above) who are not taking uric acid-lowering drugs, patients with gout who are not taking uric acid-lowering drugs
  Interventions: Dietary Supplement: Give the Placebo and test article

INTERVENTIONS:
Dietary Supplement: Give the Placebo and test article — Phase 1: The subjects take 2 capsules (500 mg/capsule)/Placebo after dinner every day for 14 days.
  Phase 2: The subjects take 2 capsules (500 mg/capsule)/test article after dinner every day for 28 days.

SUMMARY:
This study aims to investigate the efficacy of the lactic acid bacteria "LUA probiotics" in reducing serum uric acid levels. The use of health supplements prior to the onset of gout symptoms is proposed as a preventive strategy to mitigate the development of gout and to reduce the subsequent reliance on long-term pharmacological treatments. Hyperuricemia is the presence of abnormally high levels of uric acid in the blood serum. Long-term hyperuricemia is a major factor in causing gout. In addition, hyperuricemia is associated with many diseases. Therefore, the prevention and treatment of hyperuricemia has gradually attracted attention. In recent years, studies have pointed out that whether from cell experiments or animal experiments, lactic acid bacteria (LAB) have the effect of lowering uric acid. However, there is a lack of rigorous clinical observational studies to further explore whether lactic acid bacteria really have the effect of lowering uric acid. This product "LUA Probiotics" is a probiotic developed and produced by the Longtan Branch of Grape King Biotechnology Co., Ltd. Its main ingredients include Lactobacillus reuteri (Lactobacillus reuteri), β-carotene, silicon dioxide and magnesium stearate. This product is not yet commercially available.

DETAILED DESCRIPTION:
This study aims to investigate the efficacy of the lactic acid bacteria "LUA probiotics" in reducing serum uric acid levels. The use of health supplements prior to the onset of gout symptoms is proposed as a preventive strategy to mitigate the development of gout and to reduce the subsequent reliance on long-term pharmacological treatments. In recent years, lactic acid bacteria have gradually been recognized to have many benefits for human health, especially in regulating intestinal flora, enhancing immune function, and improving metabolism. Uric acid is a product of purine metabolism in the human body. Excessive uric acid concentration can cause hyperuricemia, which in turn increases the risk of gout attacks. The formation of hyperuricemia is related to multiple factors, including poor eating habits, genetic factors, and metabolic disorders.

As research on intestinal microbiota deepens, scientists have discovered that changes in intestinal flora may have a certain impact on metabolic diseases, including hyperuricemia. As an important type of probiotics, lactic acid bacteria have the ability to improve the structure of intestinal flora, regulate immune response and have anti-inflammatory effects. Recent studies have shown that lactic acid bacteria may play a positive role in reducing uric acid concentration in the blood through various mechanisms, such as degrading purine substances in the intestine, promoting uric acid excretion, and inhibiting uric acid production .

In addition, the function of lactic acid bacteria in regulating the intestinal environment, improving the diversity of intestinal microorganisms and promoting the growth of beneficial bacteria may also indirectly affect the metabolic process of uric acid. Therefore, exploring the potential of lactic acid bacteria in regulating uric acid concentration has become a hot topic in many current studies. These studies not only provide new insights into the health effects of lactic acid bacteria, but also provide new directions for the prevention and treatment of gout and other diseases related to abnormal uric acid.

This study will explore the potential role and mechanism of lactic acid bacteria in lowering uric acid and evaluate its feasibility as an adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Collect 20 people, both male and female, aged 20 or above.
2. Be conscious, willing to participate in the clinical observational research project, and complete the signed written consent form.
3. Patients with hyperuricemia (uric acid level above 7.5 mg/dL) who have not taken uric acid-lowering drugs, and patients with gout who have not taken uric acid-lowering drugs, regardless of gender.

Exclusion Criteria:

1. Patients diagnosed by a physician as suffering from a major injury or illness listed by the National Health Insurance Administration.
2. Pregnant women or women who plan to become pregnant within six months.
3. Patients with abnormal liver function (AST, ALT greater than 2 times the upper limit of normal).
4. Patients with abnormal renal function (serum creatinine > 1.5 mg/dL).
5. Patients with gastrointestinal dysfunction (surgery, frequent diarrhea).
6. Those who must continue to take antibiotics, histamine-2 antagonists, proton pump inhibitors, antioxidants, probiotics, laxatives and other drugs.
7. Patients with serious complications such as stroke, myocardial infarction, or major trauma or surgery in the past six months.
8. People who are allergic to Lactobacillus.
9. Subjects who are unable to exercise their right to consent on their own.
10. Those who have irregular eating habits and are unable to cooperate with the plan implementation.
11. Those who have poor compliance with doctor's orders.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Collect 20 people, both male and female, aged 20 or above.
  2. Be conscious, willing to participate in the clinical observational research project, and complete the signed written consent form.
  3. Patients with hyperuricemia (uric acid level above 7.5 mg/dL) who have not taken uric acid-lowering drugs, and patients with gout who have not taken uric acid-lowering drugs, regardless of gender.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
The 20 subjects should be detected the value of uric acid (mg/dL), glucose ac (mg/dL), TG (mg/dL), TC (mg/dL), HDL (mg/dL) and LDL (mg/dL). | Phase 1: The 20 subjects take 2 capsules (500 mg/capsule)/Placebo after dinner every day for 14 days. Phase 2: The same 20 subjects take 2 capsules (500 mg/capsule)/test article after dinner every day for 28 days.
  This study aims to evaluate whether taking lactic acid bacteria "LUA probiotics" can reduce blood uric acid levels, and prevent gout symptoms by taking health foods before they occur, avoiding the need to take medication later.

SECONDARY OUTCOMES:
The 20 subjects should be detected the value of uric acid (mg/dL), glucose ac (mg/dL), TG (mg/dL), TC (mg/dL), HDL (mg/dL), LDL (mg/dL), hematology (14 items) and 8 kinds of cytokine: IL-1β, IL-6, IL-10, IL-13, IL-17, IL-18, TNF-α, IFN-γ (Unit: pg/mL). | Phase 1: The 20 subjects take 2 capsules (500 mg/capsule)/Placebo after dinner every day for 14 days. Phase 2: The same 20 subjects take 2 capsules (500 mg/capsule)/test article after dinner every day for 28 days.
  This study aims to evaluate whether taking lactic acid bacteria "LUA probiotics" can reduce blood uric acid levels, and prevent gout symptoms by taking health foods before they occur, avoiding the need to take medication later.

CONTACTS AND LOCATIONS:
Overall Officials: Min-Chih Hsu, Master, Principal Investigator — Super Laboratory Co., Ltd.
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cheng S, Shan L, You Z, Xia Y, Zhao Y, Zhang H, Zhao Z. Dietary patterns, uric acid levels, and hyperuricemia: a systematic review and meta-analysis. Food Funct. 2023 Aug 29;14(17):7853-7868. doi: 10.1039/d3fo02004e. PMID 37599588